CLINICAL TRIAL: NCT00682383
Title: Phase II Trial of Combined Modality Therapy With Growth Factor Support in Locally Advanced NSCLC
Brief Title: Combined Modality Therapy With Growth Factor Support in Locally Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Rogerio Lilenbaum, M.D., Principal Investigator Rogerio Lilenbaum, M.D., Mt. Sinai Medical Center, Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LUN 07
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Unresectable Locally Advanced NSCLC
Keywords: Advanced NSCLC; Lung Cancer; Mount Sinai Medical Center CCOP
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Etoposide; Radiotherapy; Docetaxel; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARM 1 (Other): Cisplatin 75 mg/m2 day 1 and 22
  Etoposide 80mg/m2 days 1-3, 22-24
  Radiation therapy: (initial fields 1.8gy/day (5 weeks) to 45Gy, then boost 2.0Gy/day (8 days) to a total of 61Gy) beginning day 1 (Total elapsed time: approximately 6 weeks, 3 days)
  Filgrastim 5µg/kg* SQ injection days 4-13 and days 25-34
  Docetaxel 75mg/m2 Q 3 Weeks X 3 Cycles
  Pegfilgrastim 6 mg SQ injection day 2 of each cycle
  Interventions: Drug: Cisplatin; Etoposide; Radiation therapy; Docetaxel; Neulasta

INTERVENTIONS:
Drug: Cisplatin; Etoposide; Radiation therapy; Docetaxel; Neulasta — Cisplatin 75 mg/m2 day 1 and 22
  Etoposide 80mg/m2 days 1-3, 22-24
  Radiation therapy: (initial fields 1.8gy/day (5 weeks) to 45Gy, then boost 2.0Gy/day (8 days) to a total of 61Gy) beginning day 1 (Total elapsed time: approximately 6 weeks, 3 days)
  Filgrastim 5µg/kg* SQ injection days 4-13 and days 25-34
  Docetaxel 75mg/m2 Q 3 Weeks X 3 Cycles
  Pegfilgrastim 6 mg SQ injection day 2 of each cycle

SUMMARY:
To determine the safety and efficacy of administering filgrastim with concurrent chemoradiotherapy and the potential benefit of administering pegfilgrastim with consolidation chemotherapy in patients with unresectable locally advanced NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC: Either histologic or cytologic proof of a newly diagnosed non-small cell lung cancer is required. A biopsy with histology is preferred, but cytology is allowed. Histology or cytology from involved mediastinal or supraclavicular lymph nodes alone will be allowed if a separate distal primary lesion is clearly evident on radiographs (i.e., a second biopsy will not be required).
* Patients with two or more parenchymal lesions on same or opposite sides of the lung are ineligible.
* Must have unresectable Stage IIIA (N2) or IIIB disease and also satisfy the following criteria:
* Unresectable Stage IIIA (N2) patients:

  * N2 mediastinal lymph nodes must be multiple and/or bulky on CT scan or X-ray, such that, in the opinion of the treating investigator, the patient is not a candidate for induction chemotherapy or chemoradiotherapy followed by surgical resection.
  * N2 status must be documented by any one of the following methods:
  * Histologic or cytologic proof of N2 disease by exploratory thoracotomy, thoracoscopy, mediastinoscopy, mediastinotomy, Wang needle biopsy, fine needle aspiration under bronchoscopic or CT guidance or other method
  * Node positivity by PET scan
  * Nodes >2 cm on CT scan
  * Paralyzed left true vocal cord with separate left lung primary distinct from AP window nodes on CT Scan
* Stage IIIB patients:
* Pathologic documented or radiographically documented positive N3 nodes.
* Patients with positive supraclavicular or scalene lymph nodes must not have disease extending up into the cervical region evidenced by one of the following:

  * Fine needle aspiration, core needle biopsy or excisional biopsy of supraclavicular N3 nodes
  * Biopsy of contralateral mediastinal N3 nodes by mediastinoscopy, mediastinotomy, or thoracotomy
  * Fine needle aspiration, core needle or Wang needle biopsy under CT or bronchoscopic fluoroscopic guidance of enlarged contralateral N3 mediastinal nodes
  * Contralateral mediastinal nodes >2 cm on CT scan
  * Contralateral node positivity on PET scan
  * Right sided primary with paralyzed left true vocal cord
* Any of the following T4 lesions: Tumor of any size that invades any of the following: mediastinum, heart, great vessels, trachea, esophagus, vertebral body or carina:

  * Written documentation of type of T4 extent by attending surgeon if the patient has had an exploratory thoracotomy or thoracoscopy
  * T4 involvement of the trachea or carina by direct bronchoscopic visualization
  * T4 involvement of the heart, esophagus, aorta, or vertebral body documented by CT scan, MRI or transesophageal ultrasound
  * T4 involvement of the mediastinum may also be accepted by CT or MRI criteria if, in absence of the above organ involvement, there is a soft tissue extension directly into the mediastinal space.
* Radiographic criteria for involvement of main pulmonary artery or vein is allowed only if there is a mediastinal soft tissue mass.
* Age > 18 years
* ECOG performance status 0 or 1
* Ability to give informed consent
* Adequate organ and marrow function as evidenced by the following peripheral blood counts or serum chemistries at study entry:

  * WBC > 4,000/µL
  * Absolute neutrophil count > 1,500/mm3
  * Platelet count > 100 x 103 cells/mm3
  * Bilirubin < 1.5 x institutional ULN
  * AST or ALT < 2.5 x institutional ULN
  * Alkaline Phosphatase <2.5 x institutional ULN
  * Serum Creatinine < 2.0mg/dL and/or adequate creatinine clearance
* Adequate pulmonary function (FEV>1.5 liters, or if <1.5 liters, the predicted FEV1of the contralateral lung must be >800 cc based on the quantitative split function testing. (Predicted FEV1= FEV1 x % perfusion to uninvolved lung from quantitative lung V/Q scan report)
* Must have one measurable lesion by chest X-ray or CT scan. Lesion(s) must be accurately measured in at least one dimension (longest diameter to be recorded) as >20mm with conventional techniques or as >10mm with spiral CT scan
* Men and women of childbearing potential must agree to use effective contraception while on treatment and for 6 months after treatment

Exclusion Criteria:

* Malignant pleural or pericardial effusion
* Prior chemotherapy or radiation therapy
* Pregnant or lactating females
* Primary malignancy other than basal or squamous carcinoma of the skin or carcinoma in situ of the cervix, or any other cancer for which the patient has been disease free for five years. Other in situ malignancies (e.g. breast, bladder, etc) in the past 3 years are permissible
* Unintentional weight loss >10% body weight within the last 3 months
* Unable to provide informed consent
* Any pre-malignant myeloid condition or any malignancy with myeloid characteristics
* Active infection
* Known hypersensitivity to E. coli-derived proteins, pegfilgrastim, Filgrastim, or any other component of the product
* Significant nonmalignant disease including: documented HIV infection; uncontrolled heart disease, and poorly controlled diabetes
* Treatment within the last 30 days with any experimental agent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety and efficacy of administering pegfilgrastim with concurrent chemoradiotherapy and the potential benefit of administering pegfilgramstim with consolidation chemotherapy in patients with unresectable locally advanced NSCLC patients. | One year

SECONDARY OUTCOMES:
To determine the frequency of dose reductions, dose delays, and dose omissions during chemoradiotherapy with filgrastim and consolidation therapy with pegfilgrastim. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Lilenbaum, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, Miami Beach, Florida, United States